CLINICAL TRIAL: NCT06166875
Title: Accuracy of Inferior Vena Cava Collapsibility Index as a Measure of Central Venous Pressure
Brief Title: Accuracy of IVCCI as a Measure of CVP
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD186/2023
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: IVC Collapsibility Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation Sample: 80 patients will be recruited as a derivation sample to calculate the regression equation
- Validation Sample: 80 patients will be recruited as a validation sample to test the performance of the equation

SUMMARY:
The primary aim of the current study is to examine the accuracy of IVCCI for measurement of CVP and to derive equation or formula to predict CVP from IVCCI.

DETAILED DESCRIPTION:
Hemodynamic monitoring is important in the management of patients in the intensive care unit (ICU) Assessment of the intravascular volume, infusion of fluids or vasoactive drugs and maintenance of an adequate systemic perfusion is essential for reduction of the risk of organ failure and/or mortality.

The use of CVP through central venous catheter is a gold standard method that is extensively used in the ICU as it reflects the filling pressure of the right ventricle (RV) and RV preload.

Central venous cannulation has significant complications such as pneumothorax, hemothorax, arterial puncture, catheter malposition, cardiac arrhythmias, venous embolism, subcutaneous hematoma, and catheter related infection, and it is difficult to use this method in an emergency situation as it requires skilled personnel.

Measurement of IVC index by bedside ultrasound is widely used to assess the intravascular volume in adult patients and has the advantage of being non-invasive, rapid, and reliable for assessing the volume status.

Besides, related measures such as IVC diameter, IVC collapsibility, and IVC to aorta (AO) diameter have been applied clinically to assess the volume status and have been related to CVP.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years.
* Sex: Both sexes.
* BMI: <35
* Patient in whom central venous cannulation is needed for management.
* Spontaneously breathing patients.

Exclusion Criteria:

* Patients with increased intra abdominal pressure.
* Patients who not able to lie supine.
* Patients on mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the current study is to examine the accuracy of IVCCI for measurement of CVP and to derive equation or formula to predict CVP from IVCCI. | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Intensive Care, and Pain Management, Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt